CLINICAL TRIAL: NCT05398549
Title: Effects of Virtual Reality in Adhesive Capsulitis on Pain, Range of Motion and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/Lhr//19/2020 Sana Inyat
Record Dates: First submitted 2022-04-28; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Adhesive Capsulitis
Keywords: Virtual Reality ,Adhesive Capsulitis , Range of Motion
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Subjects in group A was treated with conventional physical therapy i.e. grade 1 and 2 mobilization and stretching exercise
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy (Active Comparator): Subjects in group A was treated with conventional physical therapy i.e. grade 1 and 2 mobilization and stretching exercise.
  Interventions: Other: Conventional Physical therapy
- Virtual reality group (Experimental): group B was treated with virtual reality stimulation given for 30 minutes per session through kinetic Xbox with sensory accelerator model no.1414.Two traditional training activities was used to improve shoulder Range of motion i.e. badminton and American baseball activity 12 times of the training Baseline treatment protocol hot pack and ultrasound was applied to both groups. Treatment duration for both groups was 30 minutes. Each subjects were receive a total 4 week protocol with 03 treatment sessions per week.
  Interventions: Other: Virtual reality group

INTERVENTIONS:
Other: Conventional Physical therapy — Subjects in group A was treated with conventional physical therapy i.e. grade 1 and 2 mobilization and stretching exercise
  Arms: Conventional physical therapy
Other: Virtual reality group — group B was treated with virtual reality stimulation given for 30 minutes per session through kinetic Xbox with sensory accelerator model no.1414. Two traditional training activities was used to improve shoulder Range of motion i.e. badminton and American baseball activity 12 times of the training.
  Arms: Virtual reality group

SUMMARY:
Adhesive capsulitis (AC) also known as frozen shoulder typically manifests to decrease range of motion (ROM) and function and increase pain in shoulder. Objective of this study is to find the effects of virtual reality (VR) in adhesive capsulitis on pain, range of motion and function to decrease pain and improve range of motion and function. The study design will be a quasi-experimental study that will be used to compare the effects of virtual reality with conventional physical therapy. Subjects with adhesive capsulitis meeting the predetermined inclusion & exclusion criteria will be divided into two groups using lottery method. Pre assessment will be done using visual analogue scale (VAS), shoulder pain and disability index (SPADI) tool and active shoulder flexion and abduction as subjective measurements. Subjects in group A will be treated with virtual reality stimulation given for 30 minutes per session through kinetic Xbox with sensory accelerator model no.1414. Two traditional training activities will be used to improve shoulder Range of motion i.e. shoulders finger ladder training activity and single curved shoulder training activity 12 times (3 rounds in each practice) of the training 1 . Patients will be required to complete standard training task by interacting with designed VR rehabilitative training games under the supervision of physical therapists and subjects in group B will be treated with conventional physical therapy i.e. grade 1 and 2 mobilization and stretching exercise. Baseline treatment protocol hot pack will be applied to both groups.

Treatment duration for both groups will be 30 minutes. Each subject will receive a total 6 week protocol with 02 treatment sessions per week. Post treatment reading will be recorded after the end of 2 nd , 4th and 6th treatment weeks. Recorded values will be analyzed for any change using SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges between 25 to 60
2. Both gender were included
3. Primary idiopathic type
4. No eyesight problems
5. Normal cognition and could follow instructions when using the system (score of 20 or more in mini mental state examination)
6. Clinically confirmed to ensure frozen shoulders through perform different physical tests i.e. speed tests, empty can test etc

Exclusion Criteria:

1. History of diabetes mellitus
2. Any history of previous upper limb fracture
3. Received steroids injection in the shoulder
4. Any history of systematic or malignant disease

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  Changes from the Baseline Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to mark their current pain level on the line. They can also be asked to mark their maximum, minimum, and average pain.
ROM Shoulder flexion (right) | 4 weeks
  Changes from the Baseline ROM range of Motion of Shoulder flexion was taken with the Help of Goniometer
ROM Shoulder flexion (left) | 4 weeks
  Changes from the Baseline ROM range of Motion of Shoulder flexion was taken with the Help of Goniometer
ROM Shoulder External rotation(right) | 4 weeks
  Changes from the Baseline ROM range of Motion of Shoulder External rotation was taken with the Help of Goniometer
ROM Shoulder External rotation(left) | 4 weeks
  Changes from the Baseline ROM range of Motion of Shoulder External rotation was taken with the Help of Goniometer
ROM Shoulder Abduction(right) | 4 weeks
  Changes from the Baseline ROM range of Motion of Shoulder Abduction was taken with the Help of Goniometer
ROM Shoulder Abduction(left) | 4 weeks
  Changes from the Baseline ROM range of Motion of Shoulder Abduction was taken with the Help of Goniometer
Shoulder Pain and Disability Index | 4 weeks
  Shoulder Pain and Disability Index (SPADI) is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with ADLs requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items. The pain scale is summed up to a total of 50 while the disability scale sums up to 80. The total SPADI score is expressed as a percentage. A score of 0 indicates best 100 indicates worst. A higher score shows more disability. In scoring SPADI, any question missed should be taken out of the total score of each subscale. i.e if 1 question is omitted in the pain section, the total score is divided by 40.

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Services Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No